CLINICAL TRIAL: NCT01427205
Title: Phase II Study of Cetuximab With or Without OSI-906, a Dual Insulin-like Growth Factor-1 Receptor and an Insulin Receptor Inhibitor, in Platinum-Refractory, Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: Phase II Study of Cetuximab With or Without OSI-906 in Head and Neck Squamous Cell Carcinoma (HNSCC)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-0680
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Squamous Cell Carcinoma; HNSCC; recurrent; metastatic; oral cavity; Cetuximab; C225; Erbitux; IMC-C225; OSI-906; Placebo; sugar pill; oropharynx; larynx; hypopharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Recurrence; Neoplasm Metastasis; Laryngeal Diseases | interventions — Cetuximab; 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A: Cetuximab + OSI-906 (Experimental): Cetuximab loading dose of 400 mg/m2 by vein (IV) then 250 mg/m2 weekly + OSI-906 150 mg orally twice a day. 21-Day Cycle.
  Interventions: Drug: Cetuximab; Drug: OSI-906
- Group B: Cetuximab + Placebo (Experimental): Cetuximab loading dose of 400 mg/m2 by vein (IV) then 250 mg/m2 weekly + Placebo orally twice a day. 21-Day Cycle.
  Interventions: Drug: Cetuximab; Other: Placebo

INTERVENTIONS:
Drug: Cetuximab — Loading dose 400 mg/m2 by vein once followed by 250 mg/m2 weekly (+/- 7 days).
  Other Names: C225; Erbitux; IMC-C225
Drug: OSI-906 — 150 mg by mouth twice a day.
  Arms: Group A: Cetuximab + OSI-906
Other: Placebo — Placebo taken by mouth twice daily.
  Other Names: sugar pill
  Arms: Group B: Cetuximab + Placebo

SUMMARY:
The goal of this clinical research study is to learn if the addition of OSI-906 to cetuximab can improve response. The safety of these drugs will also be studied.

Objectives:

Primary Objective(s): To assess progression-free survival (PFS) among patients with head and neck squamous cell carcinoma (HNSCC) treated with a combination of cetuximab plus OSI-906 and compare it with PFS among patients treated with cetuximab plus placebo.

Secondary Objective(s):

* To assess the safety and toxicity of these treatment regimens.
* To assess the efficacy of these two treatment regimens in terms of overall survival, response rate, and disease control rate
* To assess the efficacy of single agent OSI-906 following cetuximab treatment in terms of response rate and disease control rate in patients who cross-over from Arm B to receive single-agent OSI-906
* To explore blood-based and tissue biomarkers

DETAILED DESCRIPTION:
Cetuximab is designed to prevent or slow down the growth of cancer cells by blocking proteins on the cancer cell, called the epidermal growth factor receptor (EGFR).

OSI-906 is designed to prevent or slow the growth of cancer cells.

A placebo is not a drug. It looks like the study drug but is not designed to treat any disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups.

* If you are in Group 1, you will receive cetuximab and OSI-906.
* If you are in Group 2, you will receive cetuximab and a placebo.

Neither you nor the study doctor will know if you are receiving OSI-906 or the placebo. However, if needed for your safety, the study doctor will be able to find out which group you are in.

If the disease gets worse, the study doctor will find out which group you were in and you will be offered the chance to take OSI-906 alone if you were not already receiving it.

Study Drug Administration:

Each cycle is 21 days.

On Days 1, 8, and 15 of each cycle, you will receive cetuximab by vein. The first dose of cetuximab will be given over about 120 minutes. If it is well tolerated, each additional infusion will be given over about 60 minutes.

You will take OSI-906 or placebo by mouth 2 times every day about 12 hours apart (in the morning and evening).

You should take OSI-906 or placebo with food and a glass (up to 6 ½ ounces) of water. If you forget to take a dose, you can take it any time up to 6 hours before the next dose. You must not take the missed dose with the next dose on that same day or with a dose the next day. If you vomit after taking the tablet(s), the dose should be replaced only if the tablet(s) can actually be seen and counted. You should store the study drug/placebo at room temperature below 77°F.

In order to help decrease the risk of infusion reaction, you will receive Benadryl (diphenhydramine) by vein before the first dose of cetuximab. If the doctor thinks it is needed, you will receive diphenhydramine before every dose of cetuximab.

On Day 1 of each cycle, you will need to return all unused OSI-906 or placebo and the empty bottles.

Study Visits:

At every visit, you will be asked if you have had any side effects and to list any drugs you may be taking.

On Day 1 of each cycle (+/- 7 days):

* You will have a physical exam, including measurement of your weight.
* Blood (about 3 teaspoons) will be drawn for routine tests. You should not eat or drink anything (fast) for 8 hours before this blood draw.
* If the doctor thinks it is needed and you are able to become pregnant, you will have a blood (less than 1 teaspoon) or urine pregnancy test.

On Days 1, 8, and 15 of each cycle, your vital signs will be measured before and after you receive cetuximab.

Every 6 weeks (+/- 14 days):

* You will have an ECG.
* You will have a CT scan and/or MRI scan to check the status of the disease.

Length of Study:

You may continue to receive treatment as long as you are benefitting. You will be taken off study early if you experience any intolerable side effects, the disease get worse, the doctor thinks it is your best interest, or if you are unable to follow study directions.

Your participation on the study will be over once you have completed the end-of-treatment and follow-up visits.

End-of-Treatment Visit:

Within 30 days after the last dose of study drugs/placebo, you will have an end-of-treatment visit:

* You will have a physical exam, including measurement of your vital signs and weight
* You will be asked if you have had any side effects and to list any drugs you may be taking.
* Blood (about 3-4 teaspoons) will be drawn for routine tests.
* If the doctor thinks it is needed, you will have a CT scan or MRI scan to check the status of the disease.

Long Term Follow-Up:

About every 6 months from then on, you (or your family members or designees) will be asked about how you are doing and what treatments you may be receiving. This may be by phone, letter, email, or during clinic visits.

This is an investigational study. OSI-906 is not FDA approved or commercially available. At this time, OSI-906 is only being used in research. Cetuximab is FDA approved and commercially available for the treatment of colorectal and head/ neck cancer. The combination of OSI-906 and cetuximab is investigational.

Up to 66 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed recurrent or metastatic head and neck squamous cell carcinoma of the oral cavity, oropharynx, larynx or hypopharynx.
2. Patients must be willing to have a biopsy of tumor tissue for biomarker analysis.
3. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >/= 20 mm with conventional techniques or as >/= 10 mm with spiral computed tomography (CT) scan or magnetic resonance imaging (MRI). Measurable lymph nodes are required to be >/= 15 mm in size (short axis diameter). Measurable disease in previously radiated areas is acceptable as long as there has been documented progression.
4. Patients must have disease progression: 1) After platinum-based chemotherapy for recurrent/metastatic disease OR 2) Within 6 months of receiving definitive platinum-based combined modality therapy.
5. Previous treatment with cetuximab is allowed, as long as there has been a period >/= 6 months between the last cetuximab treatment and randomization
6. All prior cytotoxic therapy must have been completed at least three weeks prior to treatment on study.
7. Age >/= 18 years
8. ECOG performance status </= 2 or Karnofsky >/= 60%
9. Patients must have normal liver function as defined below: total bilirubin </= institutional upper limit of normal and aspartate aminotransferase (AST or SGOT)/alanine aminotransferase (ALT or SGPT) </= 2.5 * institutional upper limit of normal.
10. Patients - both males and females - with reproductive potential (ie, menopausal for less than 1 year and not surgically sterilized) must practice effective contraceptive measures throughout the study. Women of childbearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to registration.
11. Patients must provide verbal and written informed consent to participate in this study
12. Prior radiation treatment is acceptable as long as it has been completed one week prior to treatment on protocol.

Exclusion Criteria:

1. Patients may not be receiving any other investigational agents with anti-cancer activity.
2. Patients with known, untreated brain metastases. Patients with treated (irradiated or resected) brain metastases are eligible if treatment was completed >/= 28 days prior to study entry and if clinical neurologic function is stable.
3. History of severe allergic reactions attributed to compounds of similar chemical or biologic composition to OSI-906 or other agents used in the study.
4. QTc interval > 450 msec at baseline.
5. Concomitant drugs with a generally accepted risk of causing Torsades de Pointes
6. Congestive heart failure, New York Heart Association (NYHA) Class III or IV
7. History of arrhythmia which is symptomatic and requires treatment, or asymptomatic sustained ventricular tachycardia. Patients with atrial fibrillation controlled on medication are not excluded.
8. Fasting blood sugar > 150 mg/dl at baseline
9. Serious underlying medical condition which would impair the ability of the patient to receive protocol treatment, in the opinion of the treating physician.
10. Pregnant or breast-feeding females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From treatment initiation to progressive disease or death, up to 24 months for study period.
  PFS is time to progressive disease or death of any cause from randomization date, assessed every 6 weeks with a total study period of approximately 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: William N. William Jr., MD, Principal Investigator — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Website — http://www.mdanderson.org